CLINICAL TRIAL: NCT05396560
Title: Fecal Immunochemical Test for Post-polypectomy Surveillance to Reduce Unnecessary eNdoscopy (FIT2RUN Study)
Brief Title: Fecal Immunochemical Test for Post-polypectomy Surveillance to Reduce Unnecessary eNdoscopy
Acronym: FIT2RUN
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: FIT2RUN01
Record Dates: First submitted 2022-05-16; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study in a clinical setting to estimate the prevalence of advanced colorectal neoplasia (ACN) at colonoscopy in those with a history of low or high risk polyps or a family history of CRC/polyps and to verify the test performance characteristics of FIT in these populations. Using this information, a risk prediction model will be developed to help guide the choice between FIT and colonoscopy in the ongoing surveillance or screening of patients.

DETAILED DESCRIPTION:
Colonoscopy is an effective tool in reducing colorectal cancer (CRC) incidence, however, it is a limited resource that is not without risk. The overall goal of this study is to determine if Fecal Immunochemical Tests (FIT) could be an effective alternative to colonoscopy for the surveillance of patients at increased risk for CRC. The rationale for this project is that colonoscopy is both a more expensive (30-40X) and more limited resource than FIT, which because of its pivotal role in the investigation and management of many gastrointestinal conditions is constantly in demand.

Routine post-polypectomy surveillance is placing a rapidly growing demand on existing colonoscopy resources, driven in part by the rapid expansion of CRC screening programs.(1) Currently, there are not strong contemporary data to guide the use of colonoscopy or alternative tests for the surveillance of patients after the removal of low or high risk polyps, but colonoscopy is routinely recommended by screening guidelines, as historically no other reasonable options existed. Colonoscopy screening is also the default recommendation for individuals with a family history of CRC or polyps.

It is proposed that the highly sensitive and low cost FIT could replace colonoscopy for post-polypectomy surveillance and primary screening in at least some patients and, thereby, reduce costs while improving access to colonoscopy for other patients.

The following knowledge gaps must be filled prior to advocating the use of FIT for post-polypectomy surveillance or primary screening:

1. Contemporary data is lacking on the prevalence of advanced and non-advanced colorectal neoplasia at colonoscopy in a cohort of individuals with well characterized index pathology and/or family history of CRC/polyps.
2. There is limited data on the sensitivity and specificity of FIT for the detection of advanced colorectal neoplasia in these settings.
3. The factors that predict a higher risk of advanced colorectal neoplasia in those undergoing for post-polypectomy surveillance or a family history are unknown.

This is an observational study conducted in a clinical setting to estimate the prevalence of advanced colorectal neoplasia (ACN) at colonoscopy in those with a history of low or high risk polyps or a family history of CRC/polyps and to verify the test performance characteristics of FIT in these populations. Using this information, a risk prediction model will be developed to help guide the choice between FIT and colonoscopy in the ongoing surveillance or screening of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women age ≤ 74 years of age.
2. At least one risk factor for CRC that would generally lead to colonoscopy screening:

   1. Personal history of low risk polyps
   2. Personal history of high risk polyps
   3. Family history of CRC or polyps

Exclusion Criteria:

1. Known acromegaly, cystic fibrosis or high risk profession (firefighter)
2. Referred for colonoscopy due to a positive fecal immunochemical test or CT colonography
3. Known or suspected gene carrier for a familial cancer syndrome.
4. Does not meet medical criteria for colonoscopy at the CCSC.
5. Colonoscopy within the previous 30 months
6. Unable to provide written informed consent or complete questionnaires due to language barrier or other reasons.

Ages: 18 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will include eligible individuals referred to CCSC due to a personal history of low or high risk polyps and/or a family history of CRC/polyps who are medically fit and eligible to undergo colonoscopy at the Centre
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Advanced Colorectal Neoplasia (ACN) Prevalence | At time of colonoscopy
  ACN: Colorectal cancer or an advanced adenoma (> 1 cm, villous features, high grade dysplasia) or serrated polyp (> 1 cm or any conventional dysplasia).
Fecal Immunochemical Test Sensitivity and Specificity | FIT test to be completed between 3-42 days prior to participant colonoscopy
  Single fecal sample for measurement of hemoglobin using the OC-Sensor FIT. Positive if measured hemoglobin is ≥100 ng/ml (manufacturers recommended cut off).
  Sensitivity = proportion of individuals with at least one ACN who had a positive FIT.
  Specificity = proportion of individuals without advanced lesions who had a negative FIT.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hilsden, MD PhD, Principal Investigator — University of Calgary
Locations (1):
- Forzani & Macphail Colon Cancer Screening Centre, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided